CLINICAL TRIAL: NCT04560985
Title: Clinical Evaluation of Retention for Hydrophilic and Hydrophobic Resin-Based Sealants in Uncooperative Children: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Retention for Hydrophilic and Hydrophobic Sealants in Uncooperative Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Hussein A. Alharthy, Postgraduate student, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29-04-20
Record Dates: First submitted 2020-09-05; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Sound Newly Erupted First Permanent Molars With Deep Fissures Susceptible to Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrophilic sealant (Experimental): UltraSeal XT hydro™ sealant ®
  Interventions: Other: Hydrophilic fissure sealant
- Hydrophobic sealant (Active Comparator): Helioseal-F Sealant ®
  Interventions: Other: Hydrophobic fissure sealant

INTERVENTIONS:
Other: Hydrophilic fissure sealant — Hydrophilic fissure sealant on first molars
  Arms: Hydrophilic sealant
Other: Hydrophobic fissure sealant — Hydrophobic fissure sealant on first molars
  Arms: Hydrophobic sealant

SUMMARY:
To evaluate and compare the retention and cariostatic effect of hydrophilic and hydrophobic resin-based sealants for sealing pits and fissures of permanent molars in uncooperative children.

ELIGIBILITY:
Inclusion Criteria:

1. Children with good health and without any systematic diseases history which may interfere with their oral hygiene.
2. Children ranging in age from 6 to 9 years.
3. Children with bilateral fully erupted mandibular first permanent molars with deep fissures having a score of 0 following the International Caries Detection and Assessment System II (ICDAS II).
4. Uncooperative children with "definitely negative" or "negative" behavioral ratings according to the Frankl behavior classification scale.
5. Informed consent to the child's participation in the study signed by one of his/her parents/guardian.
6. No children will be excluded on the basis of gender, race, social or economic status

Exclusion Criteria:

1. Children with systemic diseases.
2. Children with oral habits affecting occlusion.
3. Children with any physical or mental disorders.
4. Children with cavitated, defected, missed or restored contralateral tooth.
5. Children with history of allergy to resin or latex.
6. Teeth with restorations, cavitated lesion, hypoplasia and any developmental defects.
7. Not approving to sign the consent.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Sealant retention scoring using Color, Coverage and Caries (CCC) system | At 3 months
Sealant retention scoring using Color, Coverage and Caries (CCC) system | At 6 months
Sealant retention scoring using Color, Coverage and Caries (CCC) system | At 12 months
Sealant retention scoring using Color, Coverage and Caries (CCC) system | At 18 months
Sealant retention scoring using Color, Coverage and Caries (CCC) system | At 24 months
Sealant retention scoring using Color, Coverage and Caries (CCC) system | At 36 months

SECONDARY OUTCOMES:
Caries scoring using Color, Coverage and Caries (CCC) system | At 3 months
Caries scoring using Color, Coverage and Caries (CCC) system | At 6 months
Caries scoring using Color, Coverage and Caries (CCC) system | At 12 months
Caries scoring using Color, Coverage and Caries (CCC) system | At 18 months
Caries scoring using Color, Coverage and Caries (CCC) system | At 24 months
Caries scoring using Color, Coverage and Caries (CCC) system | At 36 months

IPD SHARING:
Plan to Share IPD: No